CLINICAL TRIAL: NCT06537024
Title: Replication Study to Analyze the Surgical Treatment of Proximal Humeral Fracture
Acronym: ReplPHF
Status: Completed | Type: Observational
Sponsor: University Hospital Muenster (Other)
Collaborators: Universität Münster (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. J. Christoph Katthagen, Senior Consultant, University Hospital Muenster
Other Study IDs: Replication PHF
Record Dates: First submitted 2024-07-03; First posted 2024-08-05 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-07

CONDITIONS: Proximal Humeral Fracture
MeSH Terms: conditions — Shoulder Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- LPF: patients treated with locked plate fixation
- RTSA: reverse total shoulder arthroplasty
  Interventions: Procedure: RTSA

INTERVENTIONS:
Procedure: RTSA
  Groups: RTSA

SUMMARY:
The study at hand aimed to analyze the replicability of the observed treatment effects in these studies published by Koeppe et al. and Stolberg-Stolberg et al.

DETAILED DESCRIPTION:
see Protocol

ELIGIBILITY:
Inclusion Criteria:

- all patients will be included, who had an inpatient coded treatment using LPF or RTSA

Exclusion Criteria:

* Incomplete insurance status within two years before index
* Incomplete basic information
* Age<65 years
* Missing diagnosis of PHF (ICD: S42.2) within two years before surgery
* Previous surgical treatment (RTSA, LPF or other fracture fixation)
* Coded polytrauma
* Bone tumors/ bone metastasis
* Both sides or missing information of surgery side
* COVID-19 infection during index hospitalization

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients were grouped into two treatment groups: LPF (reference group) or RTSA depending on which therapy was performed first. If RTSA and LPF were coded at the same day, patients were assigned to RTSA group. Two different analysis sets were defined as follows:
  * Short-term set: including all patients.
  * Long-term set: including all patients, which were discharged alive and had an index surgery before 2022 (to guarantee a possible follow-up time of a least one year).
Sampling Method: Non-Probability Sample
Enrollment: 32953 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
30-day mortality | 30 days
  Death from any cause during the first 30-days after surgery.
Overall survival (OS) | up to 12 years
  Time from discharge of index hospitalization to death of any case.
Major adverse events during index case | through hospital stay, an average of 16 days
  See above, only events during hospitalization
Major adverse events after discharge | up to 12 years
  Time from discharge of index hospitalization to MAE as defined above
Thromboembolic events during index | through hospital stay, an average of 16 days
  See above, only events during hospitalization
Thromboembolic events (or death) after discharge | up to 12 years
  Time from discharge of index hospitalization to a thromboembolic event or death of any case.
Surgical complications during index case | through hospital stay, an average of 16 days
  See above, only events during hospitalization
Surgical complications after discharge | up to 12 years
  Time from discharge of index hospitalization to surgical complications, with death being considered as a competing risk event.

SECONDARY OUTCOMES:
Implant-associated complication during index | through hospital stay, an average of 16 days
  See above, only events during hospitalization
Non-Implant-associated complication during index | through hospital stay, an average of 16 days
  See above, only events during hospitalization
Minor outpatient complications after discharge | up to 12 years
  Time from discharge of index hospitalization to minor outpatient complications, with death being considered as a competing risk event.

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-08): https://cdn.clinicaltrials.gov/large-docs/24/NCT06537024/Prot_SAP_000.pdf